CLINICAL TRIAL: NCT02640456
Title: Mikrobiologi Ved Para- og Retropharyngeal Absces
Brief Title: Microbiology of Para- og Retropharyngeal Abscess
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tejs Ehlers Klug (Other)
Collaborators: Hospitalsenheden Vest (Other); Aalborg University Hospital (Other); Sygehus Lillebaelt (Other); Aarhus University Hospital (Other); Statens Serum Institut (Other); University of Aarhus (Other); Odense University Hospital (Other)
Responsible Party: Sponsor-Investigator, Tejs Ehlers Klug, Consultant, associate professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Other Study IDs: 51440
Record Dates: First submitted 2015-12-15; First posted 2015-12-29 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Retropharyngeal Abscess
Keywords: retropharyngeal abscess; parapharyngeal abscess; peritonsillar abscess; bacteriology; Fusobacterium necrophorum
MeSH Terms: conditions — Retropharyngeal Abscess; Peritonsillar Abscess

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tonsillar surface swabs, pus aspirates, tonsillar tissues, sera
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Para- or retropharyngeal abscess: Patients with para- or retropharyngeal abscess.
  Interventions: Biological: Bacteriology; Procedure: Type of surgery; Biological: Biochemistry; Biological: Serology
- Neck abscess: Patients with neck abscess without relation to the pharynx or salivary glands.
  Interventions: Biological: Biochemistry

INTERVENTIONS:
Biological: Bacteriology — Tonsillar surface swabs, tonsillar tissues, and pus aspirates.
  Groups: Para- or retropharyngeal abscess
Procedure: Type of surgery — Surgical approach and complications.
  Groups: Para- or retropharyngeal abscess
Biological: Biochemistry — Amylase concentration i pus aspirates.
Biological: Serology — Levels of antibodies against selected bacteria (F. necrophorum, F. nucleatum, and Group A streptococci) in acute and convalescent sera.
  Groups: Para- or retropharyngeal abscess

SUMMARY:
The aims of the study are:

1. Explore the bacteriology of para- and retropharyngeal abscess.
2. Validate the bacterial findings by exploring antibody development against F. necrophorum, F. nucleatum and S. pyogenes.
3. Compare bacteriologic findings in concomitant peritonsillar and parapharyngeal abscesses.
4. Characterize patients with para- and retropharyngeal abscess.
5. Compare the concentration of amylase in para- and retropharyngeal abscesses and neck abscesses without relation to the pharynx or salivary glands.
6. Perform gene-sequencing of F. Necrophorum strains, and compare these with strains recovered from patients with acute tonsillitis, peritonsillar abscess, and Lemierre´s syndrome.

DETAILED DESCRIPTION:
Patients:

Sixty patients aged 18 years or older with para- or retropharyngeal abscess and 12 patients with neck abscess without relation to the pharynx or salivary glands (controls) will be included at five Danish centers. Estimated time of inclusion: Four years.

Data:

Symptoms, findings, and other relevant information will be obtained at admission. Data regarding treatment and complications will be obtained after discharge.

Samples:

1. Tonsillar surface swabs (bilaterally)
2. Pus aspirate from para- or retropharyngeal abscess
3. Pus aspirate from peritonsillar abscess, if present
4. Biopsy or the entire tonsil (bilaterally)
5. Blood samples (acute and convalescent)

Investigations:

1. Bacterial cultures from tonsillar surface swabs, pus aspirates, and tonsillar tissues.
2. Antibody development against F. necrophorum, F. nucleatum and S. pyogenes from the two sera.
3. Gene-sequencing of F. Necrophorum strains.
4. Measurement of amylase concentrations in pus aspirates.

Power calculations:

Patients needed to show significant increase in anti-F. necrophorum antibody development.

Assumptions:

1. The found anti-F. necrophorum antibody levels will be compared to previous findings in electively tonsillectomized patients (9 of 47 patients had two-fold or higher increase in anti-F. necrophorum antibody levels).
2. Level of statistical significance: P = 0.05
3. Power: 90%.
4. Part of F. necrophorum-positive para- or retropharyngeal patients WHO develop two-fold or higher anti-F. necrophorum antibody levels: 73%.
5. Part of para- or retropharyngeal patients with F. necrophorum: 20%. Number of para- or retropharyngeal patients needed: 60.

Concerning comparison of amylase concentrations between patients with para- or retropharyngeal abscess and patients with neck abscesses without relation to the pharynx or salivary glands:

Assumptions:

1. Amylase concentration > 20 U/L in 0% of controls.
2. Amylase-concentration > 20 U/L in 50% af patients with para- or retropharyngeal abscess .
3. Inclusion of controls 1:3 compared to patients with para- or retropharyngeal abscess .
4. Level of statistical significance: P = 0.05
5. Power: 90%. Number of para- or retropharyngeal patients needed: 36. Number of controls needed: 12.

ELIGIBILITY:
Inclusion Criteria:

* para- or retropharyngeal abscess

Exclusion Criteria:

* refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixty patients with para- or retropharyngeal abscess. Twelve patients with neck abscess without relation to the pharynx or salivary glands (controls).
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2016-04; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Bacterial findings in aerobic and anaerobic cultures and MALDI-TOF mass spectrometry from para- and retropharyngeal abscesses | Within eight hours of patient admission
  Prevalence of potential bacterial pathogens (F. necrophorum, F. nucleatum, Prevotella species, Group A streptococcus, Group C/G streptococcus (large colony forming), S. aureus, H. influenzae, and Viridans streptococci) recovered from aerobic and anaerobic bacterial cultures from pus aspirates.

SECONDARY OUTCOMES:
Antibody Development against F. necrophorum, F. nucleatum, and S. pyogenes in patients with para- and retropharyngeal abscess | Within eight hours of patient admission (serum 1) and two to four weeks after admission (serum 2)
  Prevalence of patients with antibody development (at least two-fold increase of antibody level) against selected bacteria (F. necrophorum, F. nucleatum, and Group A streptococci)
Amylase concentrations in para- and retropharyngeal abscesses vs neck abscesses without relation to the pharynx or salivary glands | Within eight hours of patient admission.
  Comparison of amylase concentration i pus aspirates between patients with para- and retropharyngeal abscess versus patients with neck abscess not related to the pharynx or salivary glands (controls).
Comparison of bacterial recoveries in aerobic and anaerobic cultures from patients with concomitant peritonsillar and para-retropharyngeal abscess. | Within eight hours of patient admission.
  Comparison of prevalence of potential bacterial pathogens (F. necrophorum, F. nucleatum, Prevotella species, Group A streptococcus, Group C/G streptococcus (large colony forming), S. aureus, H. influenzae, and Viridans streptococci) recovered from aerobic and anaerobic bacterial cultures from pus aspirates between concomitant peritonsillar and para-retropharyngeal abscesses.

CONTACTS AND LOCATIONS:
Overall Officials: Tejs E Klug, MD, Study Chair — Aarhus University Hospital
Locations (5):
- Denmark (5):
  - Aalborg University Hospital, Aalborg, Aalborg
  - Aarhus University Hospital, Aarhus, Aarhus
  - Hospitalsenheden Vest, Holstebro, Holstebro
  - Odense University Hospital, Odense, Odense
  - Sygehus Lillebaelt, Vejle, Vejle